CLINICAL TRIAL: NCT06716112
Title: Mechanisms of Paired Vagus Nerve Stimulation (VNS) in Chronic Stroke: a Randomized, Blinded, Sham-controlled, Single-center Mechanistic Trial
Brief Title: Paired Vagus Nerve Stimulation Mechanisms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); The University of Texas at Dallas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 24-00751
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Chronic Stroke
MeSH Terms: interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active VNS first, then Sham VNS (Experimental): Patients will undergo two 6-week intervention blocks, receiving active VNS first and sham VNS second.
  Blocks consist of three 90-minute sessions per week with a licensed occupational therapist (OT). During these sessions, patients will perform rehabilitation training activities paired with active VNS during the first block and paired with sham VNS during the second block.
  Interventions: Device: Vagus Nerve Stimulation (VNS) Device; Device: Sham VNS Device; Behavioral: Upper Extremity Rehabilitation
- Sham VNS first, then Active VNS (Experimental): Patients will undergo two 6-week intervention blocks, receiving sham VNS first and active VNS second.
  Blocks consist of three 90-minute sessions per week with a licensed occupational therapist (OT). During these sessions, patients will perform rehabilitation training activities paired with sham VNS during the first block and paired with active VNS during the second block.
  Interventions: Device: Vagus Nerve Stimulation (VNS) Device; Device: Sham VNS Device; Behavioral: Upper Extremity Rehabilitation

INTERVENTIONS:
Device: Vagus Nerve Stimulation (VNS) Device — All patients will be implanted with the ReStore VNS device by an NYU neurosurgeon. During treatment sessions, study personnel will deliver a VNS burst at the completion of a training movement by pressing a button on a smart device, which wirelessly triggers active VNS stimulation.
Device: Sham VNS Device — All patients will be implanted with the ReStore VNS device by an NYU neurosurgeon. During treatment sessions, study personnel will deliver a VNS burst at the completion of a training movement by pressing a button on a smart device, which wirelessly triggers sham VNS stimulation.
Behavioral: Upper Extremity Rehabilitation — Rehabilitation training will be functional and activity-based, focusing on six task categories: reaching and grasping objects, gross movements with objects, flipping objects, inserting objects, self-feeding, and opening and closing containers.
  Three 90-minute training sessions per week will be administered by a licensed occupational therapist, over two six-week treatment blocks. Sessions will be paired with either active or sham VNS administration.

SUMMARY:
In this mechanistic study, 40 individuals with chronic stroke will be implanted with a small vagus nerve stimulation (VNS) device. The study will use a randomized, blinded, crossover design to deliver two conditions in six-week blocks: active VNS or sham VNS, each paired with upper extremity (UE) motor rehabilitation. Assessment visits will occur before and after each block, and will examine neural pathway strength, functional connectivity, and motor and non-motor behaviors. Investigators will test for VNS-induced changes in motor, cognitive, and affective systems, and will identify biomarkers predictive of clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* 22-79 years of age
* Unilateral supratentorial ischemic stroke that occurred ≥ 12 months prior to enrollment
* Upper extremity Fugl-Meyer Assessment score of 20 to 50
* Modified Rankin Score of 2, 3, or 4
* Meets all clinical criteria for VNS implantation as determined by the PI and clinical care team

Exclusion Criteria:

* Intracerebral hemorrhage or traumatic brain injury
* Deficits in language or attention that interfere with study participation
* Severe spasticity (Modified Ashworth > 3)
* Psychiatric disorders and/or cognitive impairments that would interfere with study participation, as assessed by medical evaluation
* Receiving any therapy (medication or otherwise) that would interfere with VNS, such as drugs that perturb neurotransmitter action (anticholinergics, adrenergic blockers, etc.)
* Presence of any other implanted electrical stimulation device
* Prior injury to vagus nerve
* Females of childbearing potential who are either pregnant, lactating, heterosexually active, or planning to become pregnant or heterosexually active during study participation; and who are not using, or will not agree to use, the following medically acceptable birth control methods:* (1) sterilization surgery for women, (2) Surgical Sterilization Implant for Women, (3) sterilization surgery for men, (4) long-acting reversible contraceptives (LARC) - implantable rod and IUD; (5) contraceptive shot/injection every 3 months; (6) oral contraceptives ("The Pill"); (7) contraceptive patch; and (8) vaginal contraceptive ring.
* Concurrent participation in another interventional clinical trial
* Ferromagnetic metal in head (except dental work) or torso
* Persons with a current or past: (a) medical (psychiatric, non-psychiatric) condition, disease, disorder, injury, or disability*; or (b) non-medical situation or circumstance that, in the opinion of the principal investigator, study participation: may pose a significant or undue risk to the person; make it unlikely the person will complete all the study requirements per protocol; or may adversely impact the integrity of the data or the validity of the study results. [*Examples include, but are not limited to, the following types of conditions, diseases or disorders: renal, peripheral vascular, cardiac, endocrinologic (e.g., diabetes), immunologic, psychiatric (e.g., substance use), neurologic (e.g., cognitive), or dysphagia]
* Persons with a neck circumference larger than 18.5 inches
* As determined by the principal investigator, is under current incarceration or legal detention

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Percent change in Ipsilesional CST MEP Size after Active VNS | Pre-Active VNS Treatment Block (Week 0 [Arm 1] or Week 6 [Arm 2]), Post-Active VNS Treatment Block (Week 6 [Arm 1] or Week 12 [Arm 2])
  Ipsilesional corticospinal tract (CST) motor evoked potential (MEP) size measured before and after the treatment block.
Percent change in Ipsilesional CST MEP Size after Sham VNS | Pre-Sham VNS Treatment Block (Week 0 [Arm 2] or Week 6 [Arm 1]), Post-Sham VNS Treatment Block (Week 6 [Arm 2] or Week 12 [Arm 1])
  Ipsilesional corticospinal tract (CST) motor evoked potential (MEP) size measured before and after the treatment block.

SECONDARY OUTCOMES:
Percent change in Ipsilesional CReST MEP Size after Active VNS | Pre-Active VNS Treatment Block (Week 0 [Arm 1] or Week 6 [Arm 2]), Post-Active VNS Treatment Block (Week 6 [Arm 1] or Week 12 [Arm 2])
  Ipsilesional corticoreticulospinal tract (CReST) motor evoked potential (MEP) size measured before and after the treatment block.
Percent change in Ipsilesional CReST MEP Size after Sham VNS | Pre-Sham VNS Treatment Block (Week 0 [Arm 2] or Week 6 [Arm 1]), Post-Sham VNS Treatment Block (Week 6 [Arm 2] or Week 12 [Arm 1])
  Ipsilesional corticoreticulospinal tract (CReST) motor evoked potential (MEP) size measured before and after the treatment block.
Percent Change in Arm Strength after Active VNS | Pre-Active VNS Treatment Block (Week 0 [Arm 1] or Week 6 [Arm 2]), Post-Active VNS Treatment Block (Week 6 [Arm 1] or Week 12 [Arm 2])
Percent Change in Arm Strength after Sham VNS | Pre-Sham VNS Treatment Block (Week 0 [Arm 2] or Week 6 [Arm 1]), Post-Sham VNS Treatment Block (Week 6 [Arm 2] or Week 12 [Arm 1])
Percent Change in Motor Control after Active VNS | Pre-Active VNS Treatment Block (Week 0 [Arm 1] or Week 6 [Arm 2]), Post-Active VNS Treatment Block (Week 6 [Arm 1] or Week 12 [Arm 2])
Percent Change in Motor Control after Sham VNS | Pre-Sham VNS Treatment Block (Week 0 [Arm 2] or Week 6 [Arm 1]), Post-Sham VNS Treatment Block (Week 6 [Arm 2] or Week 12 [Arm 1])
Percent Change in Individuation after Active VNS | Pre-Active VNS Treatment Block (Week 0 [Arm 1] or Week 6 [Arm 2]), Post-Active VNS Treatment Block (Week 6 [Arm 1] or Week 12 [Arm 2])
Percent Change in Individuation after Sham VNS | Pre-Sham VNS Treatment Block (Week 0 [Arm 2] or Week 6 [Arm 1]), Post-Sham VNS Treatment Block (Week 6 [Arm 2] or Week 12 [Arm 1])

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Schambra, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - The University of Texas at Dallas, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Heidi.schambra@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Heidi.schambra@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.